CLINICAL TRIAL: NCT06104241
Title: Clinical Study on the Safety and Initial Efficacy of BGT007 Cell Therapy in Patients With Recurrent/Metastatic Refractory Digestive Tract Tumors
Brief Title: BGT007 Cells for the Treatment of Refractory Digestive System Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Guangzhou Bioresette Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-BGT-007
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Cancer
Keywords: recurrent/metastatic/refractory
MeSH Terms: conditions — Gastrointestinal Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGT007 Cell Injection (Experimental): This is an exploratory study of single-arm, open, modified "3+3" dose escalation. The BGT007 cell therapy group received five progressively increased dose levels (5.0× 10^7 cells,1.0 ×10^8 cells, 3.0× 10^8 cells,1.0 × 10^9 cells,3.0 ×10^9 cells) of BGT007 cells. Each subject was observed for at least 4 weeks after cell transfusion (DLT observation period). The first two dose groups (5.0×10^7 cells and 1.0×10^8 cells) included 1 subject each, and the other three dose groups were followed by conventional "3+3" dose increments.
  Interventions: Biological: BGT007 Injection

INTERVENTIONS:
Biological: BGT007 Injection — BGT007 injection (d0) were infused intravenously once, and the dose group was 5.0× 10^7 cells,1.0 ×10^8 cells, 3.0× 10^8 cells,1.0 × 10^9 cells,3.0 ×10^9 cells.

SUMMARY:
This is an exploratory clinical study evaluating the safety and initial efficacy of BGT007 injection in the treatment of recurrent/metastatic/refractory digestive system tumors

DETAILED DESCRIPTION:
The researchers designed a single arm, open, exploratory study to improve the "3+3" dose escalation. The maximum dose or the best effective dose shall be determined according to the subject and dose increasing test to verify the safe and effective number of cells per unit weight. The improved "3+3" dose increasing design was adopted, and BGT007 cells were set with 5 dose groups that were gradually increased for treatment evaluation. The dose groups were 5.0 × 10^7cells，1.0 × 10^8cells，3.0 × 10^8cells，1.0 × 10^9cells，3.0 × 10^9cells. Cell reinfusion will be carried out on day 0 (d0), and each subject will be observed for at least 4 weeks after receiving cell reinfusion (DLT observation period).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent.
2. Age ≥18 years old, ≤70 years old, male and female.
3. Expected survival ≥ 3 months.
4. The Eastern Cancer Collaboration (ECOG) physical fitness score was 0-1.
5. Biopsy specimen or pathological wax section test (within 3 years before the signing of informed consent): Target protein test is positive.
6. At least one measurable lesion according to RECIST v1.1 solid tumor evaluation criteria.
7. Patients with recurrent/metastatic refractory digestive tract tumors (esophageal, gastric, pancreatic, or colorectal cancer) who have previously received second-line or above standard treatment failure or intolerance.
8. It is possible to establish a vein access for simple or intravenous blood collection, and there are no other contraindications for blood cell separation.
9. having adequate organ and bone marrow function, as defined below: Blood routine examination Neutrophil count (NEU #) ≥1.0×10^9/L Platelet count (PLT) ≥80×10^9/L Hemoglobin concentration ≥90g/L Liver function: subjects without liver metastases Aspartate aminotransferase (AST) ≤2.5× Upper Limit of Normal (ULN) Alanine aminotransferase (ALT) ≤2.5× Upper Limit of Normal (ULN) Total bilirubin (TBIL) ≤1.5×ULN Liver function: Subjects with liver metastases Aspartate aminotransferase (AST) ≤5× Upper limit of normal (ULN) Alanine aminotransferase (ALT) ≤5× Upper limit of normal (ULN) Liver function: Subjects with liver metastases or Gilbert syndrome Total bilirubin (TBIL) ≤2×ULN renal function Creatinine clearance (CCR) ≥50 mL/min Coagulation function International Standardized ratio (INR) ≤1.5×ULN Activated partial thromboplastin time (APTT) ≤1.5×ULN
10. Toxic side effects left over from previous anti-tumor therapy (radiotherapy, chemotherapy, targeted therapy, etc.) ≤ grade 1 (CTCAE 5.0).
11. During the study period and for 6 months after the end of dosing, fertile subjects (both male and female) must use effective medical contraception. For female subjects of reproductive age, a pregnancy test should be performed within 72 hours before the first dose and the result are negative.

Exclusion Criteria:

1. Active central nervous system metastases (except those stable after treatment).
2. HIV positive, HBsAg positive, HBV DNA copy number positive (quantitative detection ≥1000cps/ml), HCV antibody positive and HCV RNA positive.
3. Patients with mental or mental illness who cannot cooperate with treatment and efficacy evaluation.
4. Subjects with severe autoimmune diseases and long-term use of immunosuppressants.
5. Active or uncontrolled infections requiring systemic treatment during the 14 days prior to enrollment.
6. Any unstable systemic disease (including but not limited to):

   Active infections (except local infections); unstable angina pectoris; cerebral ischemia or cerebrovascular accident (within 6 months prior to screening); myocardial infarction (within 6 months before screening); Congestive heart failure (New York Heart Association [NYHA] classification ≥III); Severe arrhythmias requiring medical treatment; have a heart condition that requires treatment or uncontrolled hypertension after treatment (blood pressure > 160mmHg/100 mmHg).
7. dysfunction of important organs such as lung, brain and kidney.
8. The subject has undergone major surgery or severe trauma within 4 weeks prior to receiving cell therapy or is expected to undergo major surgery during the study period.
9. Received any systemic chemotherapy, immunotherapy, or small molecule targeted therapy within 1-2 weeks prior to an apheresis or within 5 half-lives, whichever is shorter.
10. The subject currently has or has had other malignant tumors that cannot be cured within 3 years, except cervical carcinoma in situ or basal cell carcinoma of the skin, and other malignant tumors with disease-free survival of more than 5 years.
11. Received chimeric antigen receptor modified T cells (including CAR-T, TCR-T) within six months.
12. Graft-versus-host disease (GVHD).
13. Participants who were receiving systemic steroid therapy prior to screening and who were determined by the investigator to require long-term use of systemic steroid therapy during treatment (except for inhalation or topical use); And subjects treated with systemic steroids within 72 h prior to cell transfusion (except for inhalation or topical use).
14. Severe allergies or history of allergies.
15. Subjects requiring anticoagulation therapy.
16. Pregnant or breastfeeding women, or have a pregnancy plan within six months (for both men and women)
17. Researchers believe that there are other reasons for not being included in the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT） | From day 0 to day 28
  Adverse events related to cell therapy were observed on 28 days after BGT007 injection, as specified in protocol.

SECONDARY OUTCOMES:
C max | 12 months
  The amplification of BGT007 injection in peripheral blood peaked after administration.
T max | 12 months
  Number of days of peak BGT007 injection expansion after administration.
ORR | 12 months
  Reportion of patients who achieved pre-defined tumor volume reduction and maintained the minimum time limit. Imaging examination was performed after administration, and RECIST1.1 evaluation criteria was used for evaluation.
PFS | 12 months
  The time from the onset of leukocyte apheresis to the appearance of tumor progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- he Affiliated Hospital of Xuzhou Medical University, Xuzhou, JangSu, China